CLINICAL TRIAL: NCT02565160
Title: Looking for Biomarkers in Human Joint Fluid Using Metabonomic, Microbiomic and Tribological Analysis
Brief Title: Analysis of Human Knee Joint Fluid Using Metabonomic, Genomic and Tribology Techniques
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 15/LO/0388
Record Dates: First submitted 2015-05-28; First posted 2015-10-01 (Estimated); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Osteoarthritis; Septic Arthritis; Rheumatoid Arthritis
Keywords: Osteoarthritis; Septic Arthritis
MeSH Terms: conditions — Osteoarthritis; Arthritis, Infectious; Arthritis, Rheumatoid | interventions — Arthrocentesis; Arthroplasty, Replacement

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Urine and Joint Fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Septic Arthritis: Patients suspected of having septic arthritis
  Interventions: Procedure: Intra-articular aspiration of Joint; Procedure: Joint irrigation washout; Procedure: Revision Joint Arthroplasty
- Osteoarthritis: Patients suffering with osteoarthritis undergoing an intervention
  Interventions: Procedure: Intra-articular aspiration of Joint; Procedure: Joint irrigation washout; Procedure: Total Joint Arthroplasty; Procedure: Revision Joint Arthroplasty
- Joint Revision: Patients who has a prosthetic joint in situ
  Interventions: Procedure: Intra-articular aspiration of Joint; Procedure: Revision Joint Arthroplasty

INTERVENTIONS:
Procedure: Intra-articular aspiration of Joint — Procedural sampling of the joint for diagnostic purposes
Procedure: Joint irrigation washout — Procedural washout for treatment purposes
  Groups: Osteoarthritis; Septic Arthritis
Procedure: Total Joint Arthroplasty
  Groups: Osteoarthritis
Procedure: Revision Joint Arthroplasty

SUMMARY:
Making the diagnosis underlying a painful, swollen joint currently involves aspiration followed by numerous microbiological and biochemical laboratory tests. This can be costly, time consuming and in the case of an acutely swollen joint, lead to a lengthy inpatient admission. There is an unmet need to provide a quick, easy, reliable dipstick like test to analyse joint fluid in the community, clinic, or emergency department setting.

The investigators aim to use well established metabonomic techniques to:

1. Analyse fluid from patients with swollen joints
2. Identify potential biomarkers of inflammatory, infective and osteoarthritic causes of joint swelling
3. Correlate this with lubrication and wear properties of the fluid The long term goal is to develop time saving, cost effective, non-invasive diagnostic tests to improve management of a swollen joint. The biomedical research centre at Imperial provides a unique and unparalleled clinical and scientific environment to conduct this research. The Imperial College division of Computational and Systems Medicine has an international reputation in metabonomics and this, together with the high volume of patients with swollen joints treated at Imperial National Health Service Trust (c1000/yr) ensures that the study can take place in an environment conductive to success.

DETAILED DESCRIPTION:
Swollen joints represent a diagnostic challenge. Possible diagnoses include: osteoarthritis, gout, rheumatological disease or infection. Diagnostic methods are limited to microscopy, microbiology and trace analysis. These methods can be slow, time consuming, expensive and often inconclusive.

Osteoarthritis varies in the severity of any inflammatory response and subsequent symptoms. To date no molecular link has been established to explain this ambiguity. Previous studies have identified metabolites of the inflammatory response but failed to investigate any correlation with symptoms or response to targeted injections.

Microbial infections of joints are destructive. It typically takes 2-3 days to identify a causative organism and confirm diagnosis. Recent studies suggest low-level bacterial colonisation within joints. The investigators aim to analyse the joint fluid for any bacterial colonisation using enrichment and 16S Polymerase Chain Reaction (PCR) then correlate the results to the metabolic profile. In addition the investigators aim to seek metabolites indicative of the presence of a biofilm which, if present severely limits treatment options.

Metabonomics is the quantitative measurement of the dynamic multiparametric response of a living system to pathophysiological stimuli or genetic modification. This provides a global metabolic profile despite a complex biological sample and has proven useful in many fields.

Our hypotheses are:

1. Each pathology will have a unique metabolic profile
2. Inflammatory osteoarthritis will contain a different metabolic profile and potentially biomarkers to treatment and/or response
3. Specifically the presence and detection of organism sub-type and biofilm biomarkers
4. These profiles can be characterised by analysis of blood, urine and joint fluid
5. This data can be used to generate diagnostic tests that will aid management of a swollen joint.
6. There will be a correlation between metabolic profile and lubricant properties of the joint fluid, that can be utilised in future engineering strategies to manage osteoarthritis.

1. To analyse joint fluid from osteoarthritic joints to identify potential biomarkers of the disease and further understanding of the cartilage destruction pathways 2. To assess population variances in joint fluid composition using metabonomics and whether this composition correlates to arthropathy of joints 3. To study the lubrication and wear properties of the joint fluid and understand how the metabolic profile influences lubrication and subsequently joint wear.

4. To study joint fluid using metabonomics to identify biomarkers of bacterial colonisation in tandem with microbial 16S Polymerase Chain Reaction and genomic sequencing.

Project Timeline:

Phases of the project are to be as follows:

Full research, Site and Ethical Approval: Provisional ethics is already granted. No obstacles to research and site approval are expected and this should be achieved shortly afterwards. (success = ethical approval) Expected June 2015

Sample Collection: The investigators aim to recruit 150 patients to the study capturing a conservative estimate of 10 per week. All orthopaedic patients will be targeted. The majority are expected to be recruited from the elective theatres. (success = 150 pts recruited) June - September 2015 (onwards)

Metabonomic Analysis Method Development: Establishing Nuclear Magnetic Resonance (NMR) methodology for metabolic profiling of synovial fluid as a sample matrix. Method development of Liquid Chromatography Mass Spectroscopy (LCMS) untargeted and targeted methodology for synovial fluid (success = achieving robust, sensitive methodology) October 2015

Joint Fluid Tribology: Analysis of the lubricating properties of the joint fluid (success = 150 samples assayed) October - December 2015

Metabonomic Analysis: In order to yield the maximum results the investigators aim to analyse using NMR screening with untargeted and targeted LCMS analysis. With approximately 150 patients and thus 450 body fluid samples the investigators are estimating an analysis time of 6 months (success = metabolic profiling and targeted analysis) November - April 2016

Microbial Genetic Analysis: PCR and sequencing of the microbial genetic content of the joint fluid (success = completion in 150 samples) April - June 2016

Collation of results, Analysis and Reporting: Preparation of results for submission to a journal with an impact factor >10. (success = editorial acceptance of manuscript) July - October 2016

ELIGIBILITY:
Inclusion Criteria:

* The patients will be recruited in several scenarios.

  1. Anyone receiving a diagnostic aspirate of joint.
  2. Patients undergoing joint arthroscopy
  3. Patients undergoing joint replacement
  4. Patients undergoing prosthetic joint revision surgery

Exclusion Criteria:

* No patient under 16 years or age or older than 80 years will be entered for the study.
* Any female patient who is pregnant will be excluded.
* Any patient medicated with anti-coagulants will be excluded.

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: In summary we expect to recruit 150 subjects and sample three body fluid types. In some cases control and multiple time points will be collected.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Metabolic profiling of all three body fluids in 100 + patients | 14 months

SECONDARY OUTCOMES:
DNA Profiling of 100 Joint fluid samples for the assay of the microbiome | 14 months

CONTACTS AND LOCATIONS:
Overall Officials: Chinmay Gupte, MBBChir, Principal Investigator — Imperial College London
Locations (1):
- Imperial College NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2015-01-08): https://cdn.clinicaltrials.gov/large-docs/60/NCT02565160/Prot_000.pdf